CLINICAL TRIAL: NCT02402283
Title: Comparative Randomized, Single Dose, Two-Way Crossover Open Label Bioequivalence Study of Terix Labs Ltd Metronidazole Benzoate (400 mg Metronidazole Per Sachet Oral Granules) Versus Zentiva Flagyl™ 400 mg Tablets (400 mg Metronidazole Per Film Coated Tablet), After An Oral Administration Of 400 mg to Healthy Adults Under Fasting Conditions
Brief Title: Study to Determine the Equivalence of Two Products Containing Metronidazole Benzoate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verisfield UK Ltd. Greek Branch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MET-GT007
Record Dates: First submitted 2015-03-24; First posted 2015-03-30 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Bioequivalency; two metronidazole-containing products
MeSH Terms: interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Product (Experimental): Metronidazole benzoate oral granules
  Interventions: Drug: Metronidazole benzoate oral granules
- Reference Product (Active Comparator): Flagyl 400 mg Tablets
  Interventions: Drug: Flagyl 400 mg Tablets

INTERVENTIONS:
Drug: Metronidazole benzoate oral granules — Single oral dose of 400 mg
  Arms: Test Product
Drug: Flagyl 400 mg Tablets — Single oral dose of 400 mg
  Arms: Reference Product

SUMMARY:
The purpose of this study is to determine the bioequivalence of Metronidazole benzoate (400 mg metronidazole per sachet oral granules)/Terix Labs Ltd and Flagyl™ 400 mg Tablets (400 mg metronidazole per film coated tablet)/Zentiva.

DETAILED DESCRIPTION:
This study aims to compare the absorption and disposition kinetics of two products containing metronidazole under fasting conditions. These products are: Metronidazole benzoate (400 mg metronidazole per sachet oral granules)/Terix Labs Ltd, Test product manufactured by ONE PHARMA, Greece and Flagyl™ 400 mg Tablets (400 mg metronidazole per film coated tablet)/Zentiva, a Reference product manufactured by Famar Health Care Services, Spain. The bioequivalence of a single 400 mg dose of both products will be assessed by comparing the pharmacokinetic parameters derived from the plasma concentration-time profiles for metronidazole.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years, inclusive.
* Body Mass Index (BMI) range is within 18.5 - 30 Kg/m2.
* Subject does not have a known allergy to the drug under investigation or any of its ingredients or any other related drugs.

Exclusion Criteria:

* Medical demographics performed not longer than two weeks before the initiation of the clinical study with significant deviations from the normal ranges.
* Results of laboratory tests which are outside the normal range or liver function tests (alkaline phosphatase (ALP) accepted if below reference range) that are outside the reference range or hemoglobin (Hb) or red blood cells (RBC) indices (mean corpuscular volume (MCV), MCH and mean corpuscular hemoglobin concentration (MCHC)) with deviation outside 5% of the reference range. (Laboratory tests are performed not longer than two weeks before the initiation of the clinical study).
* Acute infection within one week preceding first study drug administration.
* History of drug or alcohol abuse.
* Subject is a heavy smoker (more than 10 cigarettes per day).
* Subject does not agree not to take any prescription or non-prescription drugs within the two weeks preceding the first study drug administration until donating the last sample of the study.
* Subject does not agree not to take any vitamins taken for nutritional purposes within two days before first study drug administration until donating the last sample of the study.
* Subject is on a special diet (for example subject is a vegetarian).
* Subject consumes large quantities of alcohol or beverages containing methylxanthines e.g. caffeine (coffee, tea, cola, energy drinks, chocolate etc).
* Subject does not agree not to consume any beverages or food containing alcohol 48 hours prior to study drug administration until donating the last sample in each respective period.
* Subject does not agree not to consume any beverages or food containing methyl-xanthines e.g. caffeine (coffee, tea, cola, energy drinks, chocolate etc.) 24 hours prior to the study drug administration until the end of confinement period.
* Subject does not agree not to consume any beverages or food containing grapefruit 7 days prior to first study drug administration until donating the last sample in the study.
* Subject has a history of severe diseases which have direct impact on the study.
* Participation in a bioequivalence study or in a clinical study within the last 80 days before first study drug administration.
* Subject intends to be hospitalized within 3 months after first study drug administration.
* Subjects who donated blood or its derivatives in the past 3 months or who through completion of this study would have donated more than 1250 ml in 120 days, 1500 ml in 180 days, 2000 ml in 270 days, 2500 ml of blood in 1 year.
* The subject is a pregnant or lactating female.
* Subject has a history of significant asthma, peptic or gastric ulcer, sinusitis, pharyngitis, renal disorder (impaired renal function), hepatic disorder (impaired hepatic function), cardiovascular disorder, neurological disease such as epilepsy, haematological disorders or diabetes, psychiatric, dermatologic or immunological disorders.
* Subject who have been engaged in strenuous exercise at least one day prior to dosing till the last sample of each respective period.
* Subject having at screening examination a pulse outside the normal range of 60-100 beat per minute or a body temperature outside the normal range of 36.4-37.7 ○C or a respiratory rate outside the normal range of 14-20 breath per minute or a sitting blood pressure less than 100/60 mm Hg or more than or equal to 140/90 mm Hg.
* Subject has a history of difficulties in swallowing or any gastrointestinal disease which could affect the drug absorption.
* Subject has a history of favism (glucose-6-phosphate dehydrogenase deficiency).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Plasma concentration time profiles under the curve (AUC0-t) from zero (0) hours to time (t) | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  The area under the plasma concentration versus time curve, from time zero (0) to t hours
Maximum concentration (Cmax) | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  Maximum measured plasma concentration

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  Time of the maximum measured plasma concentration. If the maximum value occurs at more than one time point, tmax is defined as the first time point with this value
Elimination rate constant (Kel) | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  Apparent first-order elimination or terminal rate constant
Terminal half life (t1/2) | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  The elimination or terminal half-life
Area Under the plasma concentration-time curve (Auc0-infinity) from zero (0) hours to infinity | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  The area under the plasma concentration versus time curve from time (0) to infinity
Number of participants with Adverse Events | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Naji Naji, B.Sc. Pharm, Study Director — International Pharmaceutical Research Center; Abdullah Hiyari, M.D., Principal Investigator — International Pharmaceutical Research Center
Locations (1):
- International Pharmaceutical Resaerch Center (IPRC), Amman, Amman Governorate, Jordan